CLINICAL TRIAL: NCT01649128
Title: Screening Models for Early Detection of Late-onset Preeclampsia With Various Markers in Low-risk Pregnancy Populations
Brief Title: Screening for Preeclampsia With Various Markers in Low-risk Pregnancy Populations
Status: Completed | Type: Observational
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, Dong Hyun Cha, professor, CHA University
Other Study IDs: PrePark
Record Dates: First submitted 2012-07-19; First posted 2012-07-25 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Preeclampsia
Keywords: preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
For the prediction of late-onset preeclampsia (PE) in low risk women, the investigators established a cut-off value for sFlt-1/PlGF ratio and evaluated the combination models of Elecys, second trimester uterine artery (UtA) doppler, and fetoplacental proteins for Down syndrome screening.

DETAILED DESCRIPTION:
A prospective study was carried on in Cha hospital. Serum samples for Down syndrome screening were assayed to estimate pregnancy-associated plasma protein-A (PAPP-A), alpha-fetoprotein , unconjugated estriol, human chorionic gonadotrophin , and inhibin-A. Women screened for Down syndrome were offered UtA Doppler at 20-24 weeks of gestation and then collected serial serum samples for sFlt-1/PlGF ratio at two time points (24-27 and 34-37 weeks' gestation).

ELIGIBILITY:
Inclusion Criteria:

* Women considered as a potential participant in this research were patients regularly visited at the prenatal care of Cha hospital in Seoul, Korea

Exclusion Criteria:

* early onset and cases not to measure the sFlt/PlGF ratio and other markers
* twin pregnancy
* Chronic hypertension
* prior history of preeclampsia
* pregestational diabetes mellitus
* gestational diabetes mellitus
* patients delivered before 35 weeks of gestation
* preeclamptic patients with onset before 35 weeks of gestation
* patients with body mass index 25kg/m2 or greater
* maternal age 40 years older

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: low risk women who had not a risk factor of preeclampsia.
Sampling Method: Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2009-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
identification of patients at risk for late-onset preeclampsia with sFlt-1/PlGF ratio | at delivery

SECONDARY OUTCOMES:
identification of patients at risk for late-onset preeclampsia with combined biochemical markers | at delivery